CLINICAL TRIAL: NCT01108952
Title: The Impact of Chemotherapy on Memory Function and the Development of Traumatic Symptoms in Children With Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Herzog Hospital (Other)
Responsible Party: Ronit Elhasid, MD, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-RE-687-CTIL
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Oncology; Trauma; Pediatric
Keywords: Chemotherapy; Memory; Methotrexate; Glucocorticoids; Trauma; pediatric oncology; traumatization
MeSH Terms: conditions — Neoplasms; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: While treatment for pediatric cancer has improved significantly over the past 40 years, the neurotoxic side-effects of the chemotherapy agents themselves are now being recognized. Two drugs suspected of having acute impact on memory performance in children are methotrexate (MTX) and steroids (GCs). In addition, new evidence suggests that this neurotoxicity might actually protect these children from traumatization.

Working hypothesis and aims: This project aims to examine the acute impact of MTX and GC chemotherapy on memory performance in children and young adults with cancer, and the subsequent impact on the development of traumatic symptoms. We hypothesize that MTX and GCs will each produce acute declines in memory performance and that children with greater reductions in memory performance will have fewer traumatic symptoms.

Methods: The investigators will recruit 45 children being treated with MTX or GCs at Dana Children's Hospital. To determine acute impact on memory, a battery of memory tests will be administered before and after a cycle of MTX and before and after a cycle of GCs. In addition, traumatic symptoms will be assessed at each post-chemotherapy evaluation point Expected results: The investigators expect poorer memory performance after MTX and after GCs and that these performance declines will correlate with lower rates of traumatic symptoms.

Importance: The immediate impact of MTX and GCs on memory is not well known, especially in children. In addition, recent findings have led us to hypothesize that chemotherapy-induced deficits in memory function would paradoxically protect these patients from the traumatization often associated with cancer and its treatment. The proposed study will test this novel hypothesis for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of acute lymphoblastic leukemia, non-Hodgkin's lymphoma, or osteosarcoma
* treatment protocol that includes at least one cycle of methotrexate or exogenous glucocorticoid
* informed consent to participate in the study, according to institutional guidelines
* fluency in Hebrew, English, or Arabic
* age 6 to 25

Exclusion Criteria:

* Cranial irradiation within the past year
* serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study
* active meningitis or seizures occurring less than a month before study enrollment

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with cancer
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Elhasid, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel